CLINICAL TRIAL: NCT01487187
Title: The Effect of Umbilical Cord Milking on Hemodynamic Status of Preterm Infants: a Randomized Controlled Trial
Brief Title: The Effect of Cord Milking on Hemodynamic Status of Preterm Infants
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Walid El-Naggar (Other)
Responsible Party: Sponsor-Investigator, Walid El-Naggar, Primary Investigator, IWK Health Centre
Organization: IWK Health Centre (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 1002554
Record Dates: First submitted 2011-11-22; First posted 2011-12-07 (Estimated); Last update posted 2017-03-09 (Actual); Status verified 2017-03

CONDITIONS: Preterm Infants
Keywords: Cord-milking; hemodynamic; preterm infants
MeSH Terms: interventions — Umbilical Cord Clamping

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- immediate umbilical cord clamping (Active Comparator): The control group will receive immediate cord clamping at birth which is the standard of care in our institution
  Interventions: Procedure: immediate umbilical cord clamping
- Milking the umbilical cord at birth (Experimental): Infants in the cord-milked group will be placed at or below the level of the placenta, and about 20 cm of the umbilical cord (or the length of cord that is accessible if less than 20 cm) will be vigorously milked towards the umbilicus three times before clamping the cord.
  Interventions: Procedure: Milking the umbilical cord at birth

INTERVENTIONS:
Procedure: Milking the umbilical cord at birth — Infants in the cord-milked group will be placed at or below the level of the placenta, and about 20 cm of the umbilical cord (or the length of cord that is accessible if less than 20 cm) will be vigorously milked towards the umbilicus three times before clamping the cord
  Other Names: Transfusion of blood from umbilical cord to the baby
  Arms: Milking the umbilical cord at birth
Procedure: immediate umbilical cord clamping — immediate cord clamping without milking as per standard practice
  Other Names: standard practice-cord clamping
  Arms: immediate umbilical cord clamping

SUMMARY:
Very preterm babies frequently develop problems with their blood circulation during the first few days after birth. These circulation problems could affect the oxygen and blood flow to their brain and lead to effects such as bleeding in the head or delayed developmental milestones later in life. Currently the care for such problems may include transfusion of intravenous fluids or blood to the baby and/or giving the baby medications that can help circulation.

The current practice at the delivery of these babies is to immediately clamp their umbilical cords after birth. Recent research studies have shown that giving more of the baby's own blood to them at birth by delayed cord clamping (waiting for clamping the cord for about 30-90 seconds) or by milking the cord, may reduce the number of blood transfusions that these babies may need later on. It may also improve their initial blood pressure and reduce the chances of bleeding in their heads.

More research is needed to prove if either delayed cord clamping or milking the cord at birth will be better in terms of improving these babies' health.

The aim of this study is to find out if adding some blood to these babies' circulation, through milking the cord at birth, could prevent or reduce the possible problems with blood circulation and the reduced blood flow to the brain that some of these babies may have after birth.

The investigators will also investigate if milking the cord at birth could improve their long-term developmental outcome.

Hypothesis: In preterm infants less than 31 weeks' gestation, milking the umbilical cord 3 times prior to clamping, compared to immediate clamping after birth will improve systemic blood flow (as assessed by improving superior vena cava flow measured by heart ultrasound in the first 24 hours after birth)

DETAILED DESCRIPTION:
Eligible mothers will be randomized prior to delivery once preterm labour is established (cervical dilatation > 4cm and preterm birth is considered inevitable or delivery is indicated for maternal or fetal indications) to either milking of the umbilical cord of their infants (intervention group) or to clamp the cord as per standard practice (currently it is the immediate cord clamping) after birth (control group). Randomization will be done in variable block sizes and will be concealed by using opaque envelopes prepared ahead of time from a randomization table. Envelopes will be opened before the time of delivery.

ELIGIBILITY:
Inclusion Criteria:Preterm infants < 31 weeks' gestation if their mothers fulfill the following inclusion criteria:

1. admitted to the hospital for at least 2 hours before delivery in preterm labor (cervical dilatation >2 cm or having premature rupture of membranes) or if a decision to induce labour has been made by treating physician for a maternal or fetal indications).
2. at 24+0 weeks - 30+6/7 weeks gestation (by best estimate based on date of last menstrual period or early ultrasound)

Exclusion Criteria:

1. monochorionic twin or any higher order multiple pregnancy
2. major fetal congenital or chromosomal anomalies
3. significant placental abruption
4. fetal anemia/transfusion
5. Rh isoimmunization
6. intent to withhold or withdraw treatment of the infant

Ages: 24 Weeks to 31 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 73 (Actual)
Dates: Start 2011-11; Primary Completion 2018-01 (Estimated); Study Completion 2018-01 (Estimated)

PRIMARY OUTCOMES:
Systemic blood flow as reflected by mean SVC flow measured by echocardiographic study at 4-6 hours after birth. | at 4-6 hours of age

SECONDARY OUTCOMES:
low SVC flow (< 40 ml/kg/min), as assessed by echocardiography | at 4-6 and 10-12 hours of age
Hypotension | during the first 48 hours of life
  Hypotension is defiined as mean blood pressure < corresponding gestational age number for > 30 minutes
Hyperbilirubinemia and peak bilirubin level recording | during first 2 weeks of age
  Hyperbilirubinemia requiring phototherapy (as per routine unit practice)
Systemic blood flow as reflected by mean SVC flow measured by echocardiographic study at 10-12 hours after birth. | at 10-12 hours of age
Number of blood transfusions during hospital stay | at 40 weeks of corrected gestational age
Intraventricular hemorrhage (IVH) | during first 2 weeks of life
  Intraventricular hemorrhage (IVH) as diagnosed by standard-practice cranial ultrasounds
Neurodevelopmental outcome | At 36 months of age

CONTACTS AND LOCATIONS:
Overall Officials: Walid I El-Naggar, MD, Principal Investigator — IWK Health Centre- Dalhousie University
Locations (1):
- IWK Health Centre, Halifax, Nova Scotia, Canada

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] El-Naggar W, McMillan D, Hussain A, Armson A, Dodds L, Warren A, Whyte R, Vincer M, Simpson CD. Neurodevelopmental outcomes of very preterm infants who received cord milking at birth: a randomized controlled trial. Eur J Pediatr. 2022 Dec;181(12):4215-4220. doi: 10.1007/s00431-022-04638-x. Epub 2022 Oct 4. PMID 36194256
- [Derived] El-Naggar W, McMillan D, Hussain A, Armson A, Warren A, Whyte R, Simpson D. The effect of umbilical cord milking on cerebral blood flow in very preterm infants: a randomized controlled study. J Perinatol. 2021 Feb;41(2):263-268. doi: 10.1038/s41372-020-00780-2. Epub 2020 Aug 11. PMID 32782323
- [Derived] El-Naggar W, Simpson D, Hussain A, Armson A, Dodds L, Warren A, Whyte R, McMillan D. Cord milking versus immediate clamping in preterm infants: a randomised controlled trial. Arch Dis Child Fetal Neonatal Ed. 2019 Mar;104(2):F145-F150. doi: 10.1136/archdischild-2018-314757. Epub 2018 Jun 14. PMID 29903720